CLINICAL TRIAL: NCT07282210
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study to Determine Efficacy and Safety of SIL-8301 in Sickle Cell Disease (SCD) Patients With a Predominantly Hemolytic Phenotype
Brief Title: Efficacy and Safety of SIL-8301 for Control of Hemolysis in a Uniform Sickle Cell Disease Endotype
Acronym: RESCUE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biossil Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIL-8301-001
Record Dates: First submitted 2025-11-13; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Sickle Cell Disease; Sickle Cell Anaemia; Sickle Cell Anemia
Keywords: senicapoc; Anemia, Hemolytic, Congenital; Anemia, Hemolytic; Anemia; Hematologic Diseases; Hemic and Lymphatic Diseases; Hemoglobinopathies; Genetic Diseases, Inborn; Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Anemia, Sickle Cell; Anaemia, Sickle Cell
MeSH Terms: conditions — Anemia, Sickle Cell; Anemia, Hemolytic, Congenital; Anemia, Hemolytic; Anemia; Hematologic Diseases; Hemic and Lymphatic Diseases; Hemoglobinopathies; Genetic Diseases, Inborn; Congenital, Hereditary, and Neonatal Diseases and Abnormalities | interventions — senicapoc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Senicapoc (SIL-8301) (Experimental): 20 mg twice daily for 4 days, followed by 10 mg once daily for up to 24 weeks
  Interventions: Drug: Senicapoc
- Placebo (Placebo Comparator): Matching placebo tablets twice daily for 4 days, followed by once daily for up to 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Senicapoc — 10 mg tablets; administered at a loading dose of 20 mg twice daily for 4 days, followed by a maintenance dose of 10 mg once daily for up to 24 weeks
  Other Names: SIL-8301
  Arms: Senicapoc (SIL-8301)
Drug: Placebo — Tablets similar in size and color; matching administration schedule
  Arms: Placebo

SUMMARY:
SIL-8301 (senicapoc) is being developed for the chronic treatment of patients with sickle cell disease in both adults and children. The purpose of this study is to compare the effects of senicapoc to placebo in patients with sickle cell disease that have had fewer than 2 acute sickle-related painful crises per year over the preceding 2 years, and have a predominantly hemolytic phenotype, defined as presence or history of at least one hemolytic complication and a baseline Hb of 9 g/dL or less, despite receiving hydroxyurea (an oral drug used for treatment of sickle cell disease) as standard of care. Participants will take senicapoc or matching placebo daily and continue on hydroxyurea as prescribed for up to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of sickle cell disease
* 16-35 years of age
* Hb ≤ 9.0 g/dL
* History of no more than 1 acute SCD-related painful crises requiring a visit to a medical facility per year within the preceding 2 years
* History of at least one hemolytic complication
* Current treatment with hydroxyurea

Exclusion Criteria:

* Receipt of senicapoc in a previous investigational study
* Current Red Blood Cell (RBC) transfusion or exchange transfusion program
* History of pulmonary hypertension
* Active cardiovascular, neurologic, endocrine, hepatic, or renal disorders
* Diagnosis of cancer (except non-melanoma skin cancer in situ, cervical cancer in situ, or breast cancer in situ) within the last 5 years
* History of liver disease

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Hb response rate | 24 Weeks
  Proportion of participants achieving an increase in Hb of > 1 g/dL from baseline

SECONDARY OUTCOMES:
Change from baseline in hemolytic markers | 24 Weeks
Proportion of participants with a Hb increase of > 2g/dL from baseline | 24 Weeks
Percent change from baseline in urine albumin-creatinine ratio (uACR) | 24 Weeks
Change from baseline in the 6-minute walk test (6mwt) | 24 Weeks
Change from baseline in participant reported quality of life assessment overall score and subscale domain scores of the Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-ME) | 24 Weeks
Change from baseline in overall score and subscale domain scores of the Participant-Reported Outcomes Measurement Information System (PROMIS) | 24 Weeks
  PROMIS-29 for adults; PROMIS Pediatric-25 for participants <18 years of age
Sickle cell disease complication rate | 24 Weeks
  Proportion of participants experiencing at least one new or worsening hemolytic complication at any time during the study
Proportion of participants with at least one category of improvement from baseline in Clinician and Patient Global Impression of Change | 24 Weeks
Frequency of acute sickle cell-related painful crises | 28 Weeks
Incidence of AEs, SAEs, and sickle cell disease related AEs | 28 Weeks